CLINICAL TRIAL: NCT06408285
Title: A Phase I Clinical Study on the Safety, Tolerance and Pharmacokinetic Characteristics of Single Dose Escalation of TQC3927 Powder for Inhalation in Healthy Adult Subjects
Brief Title: A Study of TQC3927 Powder for Inhalation in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQC3927-I-01
Record Dates: First submitted 2024-04-29; First posted 2024-05-10 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQC3927 powder for inhalation (Experimental): TQC3927 powder for inhalation is administered as a single dose
  Interventions: Drug: TQC3927 powder for inhalation
- TQC3927 powder for inhalation placebo (Placebo Comparator): TQC3927 powder for inhalation placebo is administered as a single dose
  Interventions: Drug: TQC3927 powder for inhalation placebo

INTERVENTIONS:
Drug: TQC3927 powder for inhalation — TQC3927 is a targeted inhibitor.
  Arms: TQC3927 powder for inhalation
Drug: TQC3927 powder for inhalation placebo — TQC3927 powder for inhalation placebo contains no active substance.
  Arms: TQC3927 powder for inhalation placebo

SUMMARY:
This is a dose escalation trial. The dosing regimen involves a single-dose study. This is a single-center, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability and pharmacokinetic characteristics of TQC3927 powder for inhalation in healthy adults subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily joined the study, sign informed consent form before the study and fully understand the study content;
* Healthy subjects aged between 18 and 45 years (inclusive), both male and female;
* The male subject should weigh at least 50kg, the female subject should weigh at least 45kg. And body mass index (BMI) within 19~28 kg/m2;
* Have no pregnancy plan and voluntarily take effective contraception measures from time of screening to at least 90 days after the last dose (subjects and their partners).

Exclusion Criteria:

* Participated in any clinical trial within 3 months prior to the screening period;
* Past medical history or current cardiac, breath，endocrine, metabolic, renal, hepatic, gastrointestinal, skin, infection, hematological, neurological or psychiatric diseases/abnormalities, or related chronic abnormalities, or related chronic diseases, or acute diseases, and the investigator evaluated that the subject was not suitable for the trial;
* Individuals with a history of glaucoma, functional constipation, benign prostatic hyperplasia, urinary tract obstruction, etc;
* People who have received or are planning to receive inactive or active vaccines during the 30 days prior to the screening period and the entire study period；
* Current history of active tuberculosis, bronchiectasis or other non-specific lung diseases；
* Any history of drug allergies, Individuals with a specific history of allergies or allergies；
* Smoking more than 5 cigarettes per day or using equivalent amounts of nicotine or nicotine-containing products during the 3 months Before first administration, or those who cannot stop using any tobacco-based products during the trial；
* Regular alcohol consumption within the first 6 months of screening (women drink more than 14 standard units per week and men drink more than 21 standard units per week (1 unit = 360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine) of alcohol per week during the 3 months prior to screening, or those who cannot refrain from alcohol during the trial, or those who tested positive for alcohol breath；
* History of drug or narcotics abuse or a positive result of urine drug test at screening；
* People who have abnormal and clinically significant results in vital signs, physical examination, laboratory tests, chest radiograph and abdominal ultrasound during screening period；
* Those who have special dietary requirements and cannot follow a unified diet；
* Subjects Positive for Any of Hepatitis B Virus Surface Antigen (HBsAg), Hepatitis C Virus Antibody (Anti-HCV), Human Immunodeficiency Virus Antibody (Anti-HIV), and Treponema Pallidum Antibody (Anti-TP)；
* Pregnant or lactating women or those with positive blood pregnancy test results during the screening period；
* Subjects who are still unable to use TQC3927 inhalation powder correctly after training；
* Any situation in which the investigator believes that this poses a safety risk to the subject in the trial or may interfere with the conduct of the study, or that the investigator believes that the subject may not be able to complete the study or may not be able to comply with the requirements of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Adverse events (AE) | From the use of the investigational drug until the last study visit, up to Day 9.
  The occurrence of all adverse events (AE).
Serious adverse events (SAE) | From the use of the investigational drug until the last study visit, up to Day 9.
  The occurrence of all serious adverse events (SAE).
Abnormal security check | From the use of the investigational drug until the last study visit, up to Day 9.
  The frequency, incidence, and severity of laboratory tests, vital signs, physical examinations, electrocardiogram examinations, etc.
Pharmacokinetics:Peak concentration (Cmax) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose.
  The Cmax is the maximum observed plasma concentration of study drug.
Area Under the Concentration-Time Curve From 0 to Last Observation (AUC [0-t]) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose.
  To characterize the pharmacokinetics of TQC3927 by assessment of area under the plasma concentration time curve from the first dose to a certain time point.
Area Under the Concentration-Time Curve From Zero to Infinity (AUC [0-infinity]) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose.
  To characterize the pharmacokinetics of TQC3927 by assessment of area under the plasma concentration time curve from 0 extrapolated to infinity.
Time to reach maximum (peak) plasma concentration following drug administration (Tmax) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose
  To characterize the pharmacokinetics of TQC3927 by assessment of time to reach maximum plasma concentration after single and multiple dosing
Half-life (t1/2) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose.
  Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Apparent volume of distribution(Vd/F) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose.
  Apparent volume of distribution of the TQC3927 in plasma.
Apparent clearance (CLz/F) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose.
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
End elimination rate (λz) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose.
  Derived from semi logarithmic linear regression of eliminating phase concentration points.
Residual area percentage of the TQC3927 (AUC_%Extrap) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose
  Residual area percentage of the TQC3927 in plasma
Mean residence time from zero to last measurable concentration (MRT0-t) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose.
  The average residence time from 0:00 to the last measurable concentration time point.
Mean residence time from zero to infinity (MRT0-∞) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose.
  Average residence time from 0:00 to infinity.
Accumulated excretion of drugs in urine and feces (Aecum) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose.
  Accumulated excretion of drugs in urine and feces from zero to time t.
Accumulated excretion of drugs in urine (Aeu,cum) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose.
  Accumulated excretion of drugs in urine from zero to time t.
Accumulated excretion of drugs in feces(Aef,cum) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose.
  Accumulated excretion of drugs in feces from zero to time t.
Renal clearance (CLr) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose.
  The ability of the kidneys to clear certain substances from plasma within 1 minute.
Total drug excretion ratio in urine and feces (Fe%) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose.
  The total excretion ratio of drugs in urine and feces from zero to time t.
Drug excretion ratio in urine (Fe%u) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose.
  The proportion of drug excretion in urine from zero to time t.
Drug excretion ratio in feces (Fe%f) | Single Day1: pre-dose, at 5,15,30,45 minutes,1,2,4,6,8,12,24,36,48,72 hours after-dose.
  The proportion of drug excretion in feces from zero to time t.

CONTACTS AND LOCATIONS:
Locations (1):
- China Japan Friendship Hospital, Beijing, Beijing Municipality, China